CLINICAL TRIAL: NCT05294302
Title: A Randomized Controlled Trial of eSCCIP: An eHealth Psychosocial Intervention for English and Spanish Speaking Parents of Children With Cancer
Brief Title: Testing eSCCIP: An eHealth Psychosocial Intervention for English and Spanish Speaking Parents of Children With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Children's Hospital Los Angeles (Other); University of Virginia (Other)
Responsible Party: Principal Investigator, Kimberly Canter, Senior Research Scientist, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01CA258668-01A1 (NIH)
Record Dates: First submitted 2022-02-21; First posted 2022-03-24 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Cancer
Keywords: eHealth; pediatric cancer; parents; psychosocial intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the intervention group (eSCCIP/eSCCIP-SP) or an education control condition.
Who Masked: Outcomes Assessor
Masking Description: Investigators who are not delivering the intervention and the study biostatistician will be blinded to participant assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eSCCIP/eSCCIP-SP (Active Comparator): The Electronic Surviving Cancer Competently Intervention Program (eSCCIP) is an innovative eHealth intervention that combines cognitive behavioral and family systems therapy to provide parents and caregivers of children with cancer (PCCC) with evidence-based coping skills and psychosocial support focused on the family unit. eSCCIP has three 30-minute, self-directed, online modules which feature a unique mix of original video content and interactive activities, supplemented by three telehealth follow-up sessions. A stakeholder-informed Spanish-language adaption of eSCCIP (eSCCIP-SP) has been developed and will be offered to Spanish-speaking PCCC. eSCCIP aims to reduce acute distress and symptoms of post-traumatic stress while increasing positive coping self-appraisal and use of cognitive coping skills.
  Interventions: Behavioral: eSCCIP/eSCCIP-SP
- Coping Space (Active Comparator): PCCC randomized to the patient education control condition will be given access to a website with information about psychosocial functioning, coping, and PTSS related to pediatric cancer. This website will be hosted on the same platform as the intervention, available in English and Spanish, and will consist of information modified from CopingSpace.org. CopingSpace.org is an evidence-informed website developed by Ryan's Case for Smiles, a national organization dedicated to supporting families impacted by pediatric cancer and other chronic diseases.
  Interventions: Behavioral: Coping Space

INTERVENTIONS:
Behavioral: eSCCIP/eSCCIP-SP — eSCCIP/eSCCIP-SP is a psychosocial eHealth intervention for PCCC. It consists of four self-guided, web-based modules (including an introductory module) and three telehealth sessions with a study interventionist.
  Arms: eSCCIP/eSCCIP-SP
Behavioral: Coping Space — Coping Space is a psychosocial informational website for PCCC.
  Arms: Coping Space

SUMMARY:
It is critical to provide accessible evidence-based psychosocial support to parents and caregivers of children with cancer (PCCC) in order to mitigate individual and family-level psychosocial risks. This effectiveness trial evaluates an eHealth intervention for English- and Spanish-speaking (PCCC) with study endpoints focused on decreasing negative psychosocial sequelae (acute distress, posttraumatic stress, and anxiety) and improving coping abilities (coping self-efficacy, cognitive coping strategies). The long-term goal of this research program is to sustain and disseminate an effective, scalable, high-reach, and cost-effective intervention to provide crucial support to PCCC across the pediatric cancer trajectory.

DETAILED DESCRIPTION:
The psychosocial needs and risks of children with cancer and their families are well-documented in the literature, including the increased risk of parental distress, posttraumatic stress, and anxiety. There is a critical need to provide evidence-based psychosocial care to parents and caregivers of children with cancer (PCCC), although many challenges exist regarding in-person intervention delivery. eHealth interventions represent an exciting potential opportunity to address many of the barriers to in-person intervention delivery in this population, but are not yet widely utilized in pediatric psychosocial cancer care. The COVID-19 pandemic has further illuminated the need for flexible, acceptable, and accessible eHealth psychosocial interventions.

The Electronic Surviving Cancer Competently Intervention Program (eSCCIP) is an innovative eHealth intervention for PCCC, delivered through a combination of self-guided interactive online content and telehealth follow-up with a therapist. eSCCIP aims to decrease symptoms of acute distress, anxiety, and posttraumatic stress while improving coping abilities by delivering evidence-based therapeutic content through a flexible, easily accessible eHealth tool. The intervention is delivered to one or two PCCC per family, but content is designed to apply to the whole family system. eSCCIP is grounded in principles of cognitive-behavioral and family systems therapy and is adapted from two efficacious in-person interventions for caregivers of children with cancer, the Surviving Cancer Competently Intervention Program (SCCIP) and the Surviving Cancer Competently Intervention Program - Newly Diagnosed (SCCIP-ND). eSSCIP has been rigorously developed through a stakeholder-engaged development process involving close collaboration with PCCC, content experts in pediatric oncology and eHealth, and web design and development experts. A Spanish language adaptation of eSCCIP, El Programa Electronico de Intervencion para Superar Cancer Competentemente (eSCCIP-SP), has recently been developed following a rigorous process and is now ready for testing as well. The self-guided online modules of eSCCIP/eSCCIP-SP feature a mix of didactic video content, novel multifamily video discussion groups featuring parents of children with cancer, and hands-on interactive activities. P

The objective of the proposed study is to test eSCCIP/eSCCIP-SP in a rigorous, multisite RCT compared to an education control condition. The primary study endpoint is a reduction in acute distress from baseline to post-intervention, with secondary endpoints focused on reductions in symptoms of posttraumatic stress and anxiety ,and improvements in coping self-efficacy and cognitive coping. Data will be collected at three timepoints (baseline, post-intervention, and three-month follow-up). An additional, exploratory aim will be focused on implementation strategies and potential costs and cost-savings of eSCCIP/eSCCIP-SP, laying the groundwork for future trials focused on dissemination and implementation, stepped-care models, and intervention refinement.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be the parent or primary caregiver of a child (ages 0 - 18 years old) diagnosed with cancer.
* Participants must be able to speak and read English or Spanish.
* Participants must have access to the internet through a computer or mobile device (e.g., smartphone, tablet).

Exclusion Criteria:

* PCCC are ineligible to participate if their child is not expected to live longer than six months from the time of potential recruitment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
K-6 | Up to 20 weeks
  Questionnaire to measure acute distress.

SECONDARY OUTCOMES:
Multidimensional Scale of Perceived Social Support | Up to 20 weeks
  Questionnaire to measure perceived social support from family, friends, and significant other.
The COVID-19 Exposure and Family Impact Scale (CEFIS) | Up to 20 weeks
  The CEFIS assesses the extent to which a family has experienced or been "exposed" to COVID-19 related potentially traumatic events (e.g., economic changes, illness in family) and the impact of these events on the family's functioning and wellbeing.
Coping Self-Efficacy Scale | Up to 20 weeks
  Questionnaire to measure perceived ability to cope effectively with challenging situations across three domains (use problem-focused coping, stop unpleasant emotions and thoughts, get support from friends and family).
Cognitive Emotion Regulation Questionnaire | Up to 20 weeks
  Questionnaire to identify cognitive coping strategies used after a negative event or situation. Measures nine different cognitive coping strategies.
Distress Thermometer | Up to 20 weeks
  Single-item indicator of psychosocial distress that is widely used in the oncology.
PROMIS Short Form v1.0 - Anxiety - 8a | Up to 20 weeks
  Questionnaire measuring symptoms of anxiety.
PCL-5 | Up to 20 weeks
  Questionnaire to assess for symptoms of PTSD in civilian population.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Nemours Children's Health, Delaware, Wilmington, Delaware
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data; de-identified group data may be available to qualified researchers upon request to the principal investigator.

REFERENCES:
- [Derived] Canter KS, Ritterband L, Freyer DR, Askins MA, Bava L, Loucas C, Arasteh K, You W, Kazak AE. The Electronic Surviving Cancer Competently Intervention Program-a Psychosocial Digital Health Intervention for English- and Spanish-Speaking Parents of Children With Cancer: Protocol for Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 2;12:e46339. doi: 10.2196/46339. PMID 37267038